CLINICAL TRIAL: NCT06086288
Title: Phase II, Open Label, Single Arm Study of PembrolizumAb combiNeD With Cisplatin or carbOplatin and Etoposide in Treatment naïve Advanced meRkel Cell cArcinoma (MCC) (PANDORA Trial)
Brief Title: Study of PembrolizumAb combiNeD With Cisplatin or carbOplatin and Etoposide in Treatment naïve Advanced meRkel Cell cArcinoma (MCC)
Acronym: PANDORA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-500988-12-00
Record Dates: First submitted 2023-09-26; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: Merkel Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — pembrolizumab; Etoposide; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: Pembrolizumab, Etoposide, Cisplatin or Carboplatin

INTERVENTIONS:
Drug: Pembrolizumab, Etoposide, Cisplatin or Carboplatin — Induction Phase (4 cycles, 1Cycle=3W): Pembrolizumab 200 mg + Etoposide + Cisplatin or Carboplatin; Maintenance Phase (16 Cycles, 1Cycle=6W): Pembrolizumab 400 mg

SUMMARY:
This is an open label, multicenter, phase II study evaluating the activity and safety of pembrolizumab combined with cisplatin/carboplatin and etoposide as first line treatment in patients with advanced MCC.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female subjects with histologically confirmed diagnosis of MCC, who have not received prior systemic treatment for their advanced or metastatic MCC, are at least 18 years of age on the day of signing informed consent, will be enrolled in this study.
2. Male participants:

   A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 120 days, corresponding to time needed to eliminate any study treatments (e.g. 5 terminal half-lives for pembrolizumab and/or any active comparator/combination) plus an additional 90 days (a spermatogenesis cycle) after the last dose of study treatment and refrain from donating sperm during this period.

   Female participants:
3. A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

   a. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR b. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days (corresponding to time needed to eliminate any study treatments (pembrolizumab and/or any active comparator/combination) plus 30 days (a menstruation cycle) after the last dose of study treatment.
4. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
5. Unresectable and locally advanced, relapsed or metastatic MCC stage IIIB-IV according to American Joint Committee on Cancer (AJCC) TNM Staging Classification for Merkel Cell Carcinoma (8th ed. 2017)
6. No prior systemic treatment for metastic MCC. Subjects who received adjuvant or neoadjuvant therapy are eligible if the adjuvant/neoadjuvant therapy was completed at least 12 months prior to the onset of metastatic disease.
7. Have a life expectancy of at least 3 months.
8. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
9. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
10. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
11. Have adequate organ function (protocol table 4)

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
3. Has received prior systemic anti-cancer therapy.
4. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
6. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, transitional cell carcinoma of urothelial cancer or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
9. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
10. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
12. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
13. Has an active infection requiring systemic therapy.
14. Has a known history of Human Immunodeficiency Virus (HIV) infection.
15. Has a known history of active Hepatitis B (defined as HBV DNA is detected) or known active Hepatitis C virus (defined as HCV RNA quantitative is detected) infection.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
19. Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and antitumor activity of pembrolizumab combined with cisplatin/carboplatin and etoposide as first line treatment in MCC. | 48 months
  ORR, that will be defined as the percentage of patients achieving complete response (CR) or partial response (PR) according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
To assess safety and efficacy of pembrolizumab combined with chemotherapy as first line treatment in patients with MCC | 48 months
  Incidence of Serius Adverse Events (SAE)
To assess safety and efficacy of pembrolizumab combined with chemotherapy as first line treatment in patients with MCC | 48 months
  Incidence and severity of Adverse Events (AEs) according to NCI Common Terminology criteria Adverse Event (CTCAE), version 5.0
To assess safety and efficacy of pembrolizumab combined with chemotherapy as first line treatment in patients with MCC | 48 months
  Incidence and severity of Immune-mediated Adverse Events (imAE)
To assess safety and efficacy of pembrolizumab combined with chemotherapy as first line treatment in patients with MCC | 48 months
  Overall Survival (OS) that will be measured from the date of starting therapy to the date of death by any cause
To assess safety and efficacy of pembrolizumab combined with chemotherapy as first line treatment in patients with MCC | 48 months
  Progression Free Survival (PFS) that will be measured from the date of starting therapy to the date of disease progression or death.
To assess safety and efficacy of pembrolizumab combined with chemotherapy as first line treatment in patients with MCC | 48 months
  Duration of Response (DOR) that will be measured from the date of the first response to disease progression or death in those patients who achieved a CR o PR during study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Pusceddu, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale Tumori Milano
Locations (3):
- Italy (3):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - AOUS Policlinico Le Scotte, Siena
  - Azienda Ospedaliera Universitaria Integrata (AOUI), Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oldani S, Prinzi N, Morano F, Cingarlini S, Di Giacomo AM, Niger M, Prisciandaro M, Raimondi A, Randon G, Pircher CC, Borghesani M, Valente M, Rostanzo E, Milione M, Sabella G, Cascella T, Ghelardi F, Sciortino C, Gusmaroli E, Nasca V, de Braud F, Pietrantonio F, Pusceddu S. Design and rationale of the phase II PANDORA trial: first line chemo-immunotherapy in advanced Merkel cell carcinoma. Future Oncol. 2025 Jul;21(17):2127-2133. doi: 10.1080/14796694.2025.2514402. Epub 2025 Jun 12. PMID 40501309

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT06086288/Prot_SAP_000.pdf